CLINICAL TRIAL: NCT04962139
Title: A Randomized, Double-Blind, Parallel-Group, Vehicle-Controlled, Phase-III Study to Evaluate the Safety and Efficacy of ON101 Cream for the Treatment of Chronic Diabetic Foot Ulcers
Brief Title: Evaluate the Safety and Efficacy of ON101 Cream for the Treatment of Chronic Diabetic Foot Ulcers
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to the product development strategy adjustment, the Sponsor terminated this study.
Sponsor: Oneness Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ON101CLCT04
Record Dates: First submitted 2021-07-02; First posted 2021-07-14 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Chronic Diabetic Foot Ulcers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ON101 Cream plus Standard of Care (Experimental): ON101 cream will be applied twice daily for up to 20 weeks to the Target Ulcer. The SOC will include evaluation to ensure adequate blood flow, wound cleaning, removal of necrotic, infected and/or nonviable tissue by debridement, maintenance of a moist wound environment via regular dressing changes, and management of infection through oral antibiotics, if necessary.
  Interventions: Drug: ON101 Cream
- Vehicle Cream plus Standard of Care (Placebo Comparator): Vehicle cream will be applied twice daily for up to 20 weeks to the Target Ulcer.
  The SOC will include evaluation to ensure adequate blood flow, wound cleaning, removal of necrotic, infected and/or nonviable tissue by debridement, maintenance of a moist wound environment via regular dressing changes, and management of infection through oral antibiotics, if necessary.
  Interventions: Other: Vehicle Cream

INTERVENTIONS:
Drug: ON101 Cream — Active ingredients: Extracts of Plectranthus amboinicus and Centella Asiatica
  Arms: ON101 Cream plus Standard of Care
Other: Vehicle Cream — ON101 Cream Placebo
  Arms: Vehicle Cream plus Standard of Care

SUMMARY:
The primary efficacy endpoint for this study is the proportion of subjects with complete closure of Target Ulcer during the 20-week Treatment Phase, which is assessed by the blinded independent evaluator.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects, male or female, aged 18 to 80 years (inclusive) with Type 1 or Type 2 diabetes undergoing therapy for glycemic control using available diabetes drugs including insulin.
2. Subject has a glycosylated hemoglobin, HbA1c ≦ 12%.
3. Presence of at least one diabetic foot ulcer that meets all of the following criteria:

   1. A full-thickness ulcer of UTWCS Grade I-A or II-A
   2. Ulcer size (area) is > 1 cm2 and ≤ 20 cm2 (post-debridement at time of screening and randomization)
   3. Ulcer is located on or below the malleoli and presents duration of between 6 weeks and 12 months (at time of screening).
   4. There is a minimum 3 cm margin between the qualifying Target Ulcer and any other ulcers on the specified foot (post-debridement)
   5. No active infection by clinical inspection as defined by IDSA/IWGDF criteria Note: If the subject has more than one qualifying diabetic foot ulcer, the most severe ulcer will be designated as the target ulcer.
4. Subject has adequate vascular perfusion of the affected limb, confirmed by Ankle-Brachial Index (ABI) > 0.8 and < 1.3, and transcutaneous pressure of oxygen (TcPO2) > 30 mmHg on at least one lead.
5. Subject, if female of child-bearing potential, has a negative serum pregnancy test at screening, must not be breastfeeding, and willing to use 2 medically accepted methods of contraception (e.g., barrier contraceptives [female condom, or diaphragm with a spermicidal gel], hormonal contraceptives [implants, injectables, combination oral contraceptives, transdermal patches, or contraceptive rings], and intrauterine devices) during the study (excluding women who are not of childbearing potential and/or who have been sterilized).
6. Subject should be able to walk and stand on the non-target ulcer limb.
7. Subject is willing to use an off-loading device for the target ulcer on the plantar while ambulation for the duration of the study.
8. Subject / identified caregiver trained on the study procedures is able and willing to comply with study procedures.
9. A signed and dated informed consent form has been obtained from the subject prior to any study-related procedures being performed.

Exclusion Criteria:

1. In response to standard of care, ulcer size reduction is > 30% during the two-week run-in Screening Period (between the first Screening Visit/V0 and Baseline/V2).
2. Ulcers with exposed bone or associated with osteomyelitis. Note: The osteomyelitis should be ruled out by clinical examination (probing of the wound) and X-ray findings.
3. Presence of necrosis, purulence or sinus tracts that cannot be removed by debridement.
4. Body mass index (BMI) > 42 kg/m2
5. Laboratory values at Screening of:

   1. White Blood Cells (WBC) < 3.0 X 109 cells/L；> 12.0 X 109 cells/L
   2. Liver function studies [Total bilirubin, aspartate aminotransferase (AST) and alanine transaminase (ALT)] > 3x the upper limit of normal
   3. Albumin < 2.5 g/dL
   4. Renal function studies [Serum Creatinine and Urea] > 3x the upper limit of normal
6. Presence of any clinically significant medical condition(s) in medical history during screening period that, in the opinion of the investigator, could interfere with wound healing, including but not limited to the following:

   1. Acute or unstable Charcot foot
   2. Current sepsis
   3. Active malignant disease. A subject, who has had a malignant disease in the past, was treated and is currently disease-free, may be considered for study entry.
   4. Acquired immune deficiency syndrome (AIDS) or HIV positive.
7. Subject is currently receiving (i.e., within 30 days of randomization visit) or scheduled to receive any of following medication or therapies, could interfere with wound healing during the study.

   1. immunosuppressants (including chronic systemic corticosteroids)
   2. cytotoxic chemotherapy
   3. cytostatic therapy
   4. autoimmune disease therapy
   5. dialysis
   6. lower limb revascularization surgery (e.g., angioplasty, artery bypass surgery)
   7. growth factors
   8. hyperbaric oxygen therapy
   9. bioengineered tissue or skin substitutes
   10. application of topical steroids to the ulcer
   11. use of any investigational drug(s)
8. Subjects whose non-target ulcer limb is disabled or amputated above the ankle.
9. Subject's target ulcer is located on the plantar foot with all toes amputated.
10. Subjects who need to stand continuously for more than 4 hours / day and have difficulty complying with off-loading instruction.
11. A psychiatric condition (e.g., suicidal ideation), current or chronic alcohol or drug abuse, determined from the subject's medical history, which, in the opinion of the Investigator, may pose a threat to subject compliance.
12. Has any other factor which may, in the opinion of the investigator, compromise participation and/or follow-up in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects with complete closure of Target Ulcer | 20-week Treatment Phase
  The primary efficacy endpoint for this study is the proportion of subjects with complete closure of Target Ulcer during the 20-week Treatment Phase, which is assessed by blinded independent evaluators.

SECONDARY OUTCOMES:
Time to complete closure of Target Ulcer | 20-week Treatment Phase
  Time to complete closure of Target Ulcer during the 20-week Treatment Phase, which is assessed by blinded independent evaluators.
The proportion of patients with Target Ulcer recurrence | 12-week Follow-Up Phase
  The proportion of patients with Target Ulcer recurrence during the Follow-Up Phase.
Mean change in EQ-5D-5L utility score | Day 141
  Mean change from baseline in EQ-5D-5L utility score at V12/EOT.

CONTACTS AND LOCATIONS:
Overall Officials: Shyi-Gen Chen, Study Director — Oneness Biotech Co., Ltd.
Locations (14):
- United States (14):
  - Oneness Investigational Site, Mesa, Arizona
  - Oneness Investigational Site, Carlsbad, California
  - Oneness Investigational Site, Castro Valley, California
  - Oneness Investigational Site, Fresno, California
  - Oneness Investigational Site, San Francisco, California
  - Oneness Investigational Site, Sylmar, California
  - Oneness Investigational Site, Miami, Florida
  - Oneness Investigational Site, Miami Lakes, Florida
  - Oneness Investigational Site, North Miami Beach, Florida
  - Oneness Investigational Site, Mount Prospect, Illinois
  - Oneness Investigational Site, O'Fallon, Illinois
  - Oneness Investigational Site, Springfield, Illinois
  - Oneness Investigational Site, Dallas, Texas
  - Oneness Investigational Site, McAllen, Texas